CLINICAL TRIAL: NCT05558865
Title: Evaluating the Effectiveness of a Digital Therapeutic (Somnovia) for People With Insomnia Disorder - a Randomized Controlled Trial
Brief Title: Effectiveness of a Digital Health Application for People With Insomnia Disorder (Somnovia)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: University Hospital Schleswig-Holstein (Other); University Hospital Freiburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: somnovia-RCT
Record Dates: First submitted 2022-09-26; First posted 2022-09-28 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-06

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- somnovia (Experimental): somnovia is a digital health application for people with Insomnia Disorder. Content is continuously adapted to patients' concerns and needs. somnovia is a comprehensive program, which is conceptually and substantially based on the Cognitive Behavioral Therapy for Insomnia (CBT-I) used in patients with Insomnia Disorder. It contains interactive dialogues that can be accessed via computer or smartphone, illustrations, audio recordings and motivating text messages. Techniques to cope with insomnia symptoms (e.g., psychoeducation about causes and basic emotional needs in addition to relevant strategies to improve sleep quality) are conveyed in interactive sequences that are accompanied by audio recordings, illustrations, and worksheets. Patients are also prompted to regularly complete brief symptom severity self-monitoring questionnaires. Optional daily text messages with motivational content accompany the program. The program can be accessed for 365 days after registration.
  Interventions: Behavioral: somnovia
- Care as Usual (No Intervention): Care as Usual: In the CAU control group, participants are free to continue to engage with any treatment they require. However, they will be offered access to somnovia after 6 months post-baseline.

INTERVENTIONS:
Behavioral: somnovia — Participants receive access to the digital health application somnovia
  Arms: somnovia

SUMMARY:
The trial aims to evaluate the effectiveness of a novel digital health application (somnovia), which was designed to increase sleep quality in persons with insomnia disorder. Therefore, 290 people with insomnia disorder will be recruited and randomized to two groups: (1) a control group, in which they may engage with any treatment for insomnia disorder and are offered access to somnovia after a delay of 6 months (i.e., Care-as-Usual [CAU]), or (2) to a treatment group that immediately receives 6-month access to somnovia and may also use CAU. The primary outcome measure is the score of the Insomnia Severity Index (ISI), collected at three months post-baseline.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic insomnia
* impaired quality of sleep (Insomnia Severity Index Score ≥ 10)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | 3 months after randomization
  The ISI is a 7-item patient-reported outcome measure (PROM) assessing the nature, severity, and impact of insomnia on a 5-point Likert scale to rate each item from 0 (no problem) to 4 (very severe problem).

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | 6 months after randomization
  The ISI is a 7-item patient-reported outcome measure (PROM) assessing the nature, severity, and impact of insomnia on a 5-point Likert scale to rate each item from 0 (no problem) to 4 (very severe problem).
Patient Health Questionnaire (PHQ-9) | 3 months and 6 months after randomization
  The PHQ-9 is a well-validated nine-item self-report questionnaire developed to score each of the nine DSM-IV criteria for major depressive disorder on a 4-point Likert scale, from "0" (not at all) to "3" (nearly every day).
Generalized Anxiety Disorder Assessment (GAD-7) | 3 months and 6 months after randomization
  The GAD-7 is a self-administered patient questionnaire used as a screening tool and severity measure for generalized anxiety disorder (GAD)
Work and Social Assessment Scale (WSAS) | 3 months and 6 months after randomization
  WSAS is a 5-item self-report scale to measure the ability to work in regard to physical, mental and social health as well as age group referenced competence for performance. Each item is rated on a 9-point Likert scale from 0 = "not at all impaired" to 8 = "very severely impaired".
Responder Rate on Insomnia Severity Index | 3 months after randomization
  A Responder is defined as a patient with an improvement of > 6 points on the total score of the Insomnia Severity Index from T0 to T1
Remission Rate on Insomnia Severity Index | 3 months after randomization
  Remission is defined as patients with a total score on the Insomnia Severity Index of < 8

CONTACTS AND LOCATIONS:
Overall Officials: Robert Göder, Prof. Dr., Principal Investigator — Christian-Albrechts-Universität zu Kiel, Clinic for Psychiatry and Psychotherapy
Locations (1):
- GAIA AG, Hamburg, Germany